CLINICAL TRIAL: NCT03114358
Title: A Cluster Randomized Controlled Trial Comparing Early and Late Carbapenems De-escalation in the Medicine Units, Maharaj Nakorn Chiang Mai Hospital
Brief Title: Carbapenems De-escalation as Antimicrobial Stewardship
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chiang Mai University (Other)
Responsible Party: Principal Investigator, Romanee Chaiwarith, Associate professor, Chiang Mai University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 3629
Record Dates: First submitted 2017-04-03; First posted 2017-04-14 (Actual); Last update posted 2017-04-19 (Actual); Status verified 2017-04

CONDITIONS: Anti-Bacterial Agents
Keywords: De-escalation; Carbapenems; Antimicrobial stewardship

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early carbapenems de-escalation (Experimental): De-escalation carbapenems within 24 hours or no later than 72 hours of prescription by Infectious disease specialist (early de-escalation).
  Interventions: Other: Early Carbapenem de-escalation
- Late carbapenems de-escalation (No Intervention): De-escalation followed the hospital policy in which carbapenems were evaluated by ID specialist at 72 hours of admission (late de-escalation). De-escalation may occurred earlier depends upon the decision of the primary care team

INTERVENTIONS:
Other: Early Carbapenem de-escalation — The intervention group is de-escalation carbapenems early within 24 hours or no later than 72 hours of prescription by ID specialist (early de-escalation).
  Arms: Early carbapenems de-escalation

SUMMARY:
Early de-escalation of carbapenems can reduce unnecessary use of carbaepenems compared with late de-escalation without compromised clinical outcomes

DETAILED DESCRIPTION:
A cluster randomized control trial was conducted among patients receiving care at the medicine units of the Maharaj Nakorn Chiang Mai Hospital.

Patients were randomly assigned into 2 groups. The standard group followed the hospital policy in which carbapenems were evaluated by ID specialist at 72 hours of admission (late de-escalation). De-escalation may occurred earlier depends upon the decision of the primary care team. The intervention group is de-escalation carbapenems early within 24 hours or no later than 72 hours of prescription by ID specialist (early de-escalation).

Clinical outcomes included rate of de-escalation within the first 24 hour, the mortality rate, and other clinical outcomes.

ELIGIBILITY:
Inclusion criteria

* All adult patients aged ≥ 15 years old
* received carbapenems (meropenem and imipenem/cilastatin) empirically within 24-72 hours for the first time during admission
* able to sign informed consent

Exclusion criteria

* They were in the intensive care units, or had neutropenia (absolute neutrophil count < 1,000 cell/mm3)

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2017-02-28 (Actual); Study Completion 2017-02-28 (Actual)

PRIMARY OUTCOMES:
The rate of de-escalation within the first 24 hour | 24 hours
  Compare the rate of de-escalation within the first 24 hour between arm 1 and arm 2

SECONDARY OUTCOMES:
Mortality rate | 90 days
  Compare the mortality rate between 2 groups
Readmission within 30 days, | 30 days
  Compare the rate of readmission within 30 days between 2 groups
Costs of carbapenems | 30 days
  Compare the cost of carbapenem prescription between 2 groups

IPD SHARING:
Plan to Share IPD: No